CLINICAL TRIAL: NCT04426786
Title: The Effect of Exercise on Brain Energetics in Parkinson's Disease
Brief Title: Exercise & Brain Energetics in PD
Acronym: EBEPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pacific Parkinson's Research Centre (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: H19-01839
Record Dates: First submitted 2020-06-02; First posted 2020-06-11 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Exercise; Brain energetics; Positron Emission Tomography; MRI; PET
MeSH Terms: conditions — Parkinson Disease; Motor Activity | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate intervention start: active exercise (Active Comparator): Immediately starts the six month intervention of active exercise following the baseline scan.
  Interventions: Other: Active exercise
- Delayed intervention start: passive exercise (Placebo Comparator): Starts the six month intervention of active exercise six months after the baseline scan. During the six month delay, participants in this arm undergo passive exercise.
  Interventions: Other: Active exercise; Other: Passive exercise

INTERVENTIONS:
Other: Active exercise — Thrice-weekly supervised intense aerobic exercise classes on cycle ergometers, in groups, for six months. Percentage of VO2 max will be used to regulate exercise intensity, based on an initial aerobic exercise test.
Other: Passive exercise — Thrice-weekly supervised passive exercise classes consisting of stretching and/or yoga, in groups, for six months.
  Arms: Delayed intervention start: passive exercise

SUMMARY:
There is increasing evidence that the usage and delivery of energy to the brain, known as brain energetics, is altered in people with Parkinson's disease (PD). This project will explore whether exercise has a positive impact on brain energetics using functional Magnetic Resonance Imaging (fMRI) and Positron Emission Tomography (PET) brain scanning in PD subjects.

PD subjects will be scanned before and after a supervised exercise program to investigate the effect of exercise on brain energetics. In a separate study, the investigators will also scan healthy volunteers to compare brain energetics in the healthy brain with the brain energetics data in PD subjects acquired in this study.

DETAILED DESCRIPTION:
Previous work has investigated the link between decreased brain energetics (through mitochondrial dysfunction), though an investigation in-vivo has never been feasible due to technology constraints. Furthermore, recent work has suggested exercise may help reduce the effect of mitochondrial dysfunction. There is thus compelling evidence to investigate brain energetics/mitochondrial function in-vivo, in health, at different stages of disease and the relationship to exercise. While such measurements are intrinsically difficult, a useful measure is expected to be derived from the ratio between the cerebral metabolic rate of oxygen (CMRO2) and the cerebral metabolic rate of glucose (CMRGlu), if they are measured simultaneously. The simultaneous aspect of the two measurements is extremely important as diurnal variations in CMRO2 can be as high as 20%, while those in CMRGlu as high as 38%. Fortunately, given recent advances in measurement technique and instrumentation development, such studies are now becoming possible: CMRO2 can be obtained using very advanced functional magnetic resonance imaging (fMRI) techniques with respiratory manipulations, while CMRGlu can be estimated by positron emission tomography (PET) using the tracer 18F-fluorodeoxyglucose (FDG-PET). A lower-than-normal ratio between CMRO2 and CMRGlu coupled with a decrease in CMRGlu in any brain area is taken to be indicative of locally impaired brain energetics, related to altered mitochondrial function.

The investigators hypothesize that (i) brain energetics, measured as the ratio CMRO2/CMRGlu is altered early in Parkinson's disease (PD) compared to age-matched healthy controls (HC) and continues to be altered as disease progresses; and (ii) exercise will positively affect alterations in brain energetics in PD subjects.

The investigators will recruit up to 30 PD subjects who are not habitual exercisers and up to 10 PD subjects who are habitual exercises. The 30 non-exercisers will undergo a supervised six month exercise intervention in groups, with PET/MRI scans before and after. The 10 exercisers will only be scanned once (for observational comparisons with the non-exercisers at baseline) and will not undergo the exercise intervention. In a separate study, the investigators will recruit up to 30 HCs to compare to compare their brain energetics metrics with those of the PD subjects at baseline to test hypothesis (i). Of the 30 non-exercisers, half will be assigned to start the exercise intervention immediately after their baseline scan, and the other half will have a six month delayed start to the intervention. During the delay, subjects will perform passive exercise in groups, to control for social interaction and possible placebo effects. Longitudinal comparisons of the non-exercisers before and after the intervention will test hypothesis (ii).

The objectives of this study are twofold: to (i) investigate a disease-initiating mechanism (abnormal mitochondrial function and impaired cellular bioenergetics), which could constitute a novel therapeutic target; and to (ii) study the effects of the intervention: while this will be a pilot study, involving limited exercise regimens, any knowledge gained about the impact of exercise on brain energetics will have a tremendous impact on the design of neuroprotective therapies and personalized treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Idiopathic PD according to UK Brain Bank criteria (modified to permit inclusion of subjects with a family history)
2. Mild to moderate Parkinsonism (Hoehn & Yahr stages I-III)
3. Currently exercise less than 120 minutes per week (PD non-exercisers)

General exclusion criteria:

1. atypical Parkinson syndrome (progressive supranuclear palsy, multiple system atrophy, drug-induced etc.);
2. significant osteoporosis or arthritis;
3. history of cancer within 5 years of study participation;
4. high dose of radiation from other procedures within the year;
5. not able to tolerate being off PD medication for up to 24 hours;
6. a female subject who is breast-feeding or pregnant;
7. current or past substance use problems;
8. serious head injury with loss of consciousness for ≥ 5 minutes;
9. people with other chronic diseases such as diabetes, kidney problems, high blood pressure, other known neurological disorders, or heart diseases;
10. people who report having a significant respiratory disorder (e.g. asthma, chronic obstructive pulmonary disease (COPD)) or using home oxygen will be excluded to avoid discomfort or breathing difficulties from respiratory manipulations.
11. current or past neurological disorder (e.g. strokes, seizures, neurodegenerative disease other than Parkinson's disease);
12. current or past psychiatric disorders (e.g. depression, anxiety disorders);
13. severe claustrophobia (a fear of closed in spaces);
14. weight of more than 158kg (347 lbs);
15. inability to lay still for up to 90 minutes;
16. are not medically cleared to exercise;
17. certain medications or conditions may impact participant's ability to participate and these will be discussed on a case by case basis with the participant and the study team.

MRI-specific exclusion criteria:

1. Machinist or metalworkers;
2. cardiac pacemakers, wires, or defibrillator;
3. past injury where a piece of metal lodged in your eye or orbit;
4. ferromagnetic aneurysm clip;
5. artificial heart valve;
6. electrical stimulator for nerves or bones;
7. ear or eye implant;
8. implanted drug infusion pump;
9. coil, catheter, or filter in any blood vessel;
10. orthopedic hardware (artificial joint, plate, screws);
11. other metallic prostheses;
12. shrapnel, bullets, or other metal fragments;
13. dentures, braces, or retainer;
14. surgery (brain or otherwise), tattoos, or injection into a joint in the last 6 weeks;
15. pierced body parts (other than earrings) or tattooed eyeliner;
16. non-MRI safe intrauterine device (IUD).

Subjects may be excluded following study enrollment if they meet any of the following exclusion criteria:

1. significant cognitive impairment or depression;
2. significant or unstable cardiovascular or respiratory disease - all subjects will undergo a screening aerobic exercise test;
3. failure to comply with the exercise intervention program by not completing at least 60 of the 72 exercise classes.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-26 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
PET/MRI | Six months
  CMRO2 will be computed from MRI data and CMRGlu from PET data; their ratio will be used to assess brain energetics.

OTHER OUTCOMES:
Clinical measure: motor function | Six months
  Motor function will be assessed using the MDS-Unified Parkinson's Disease Rating Scale (part III). The scale consists of 18 questions with each assigned a value in the range 0-4. Higher values indicate increasingly severe motor complications.
Clinical measure: cognitive function | Six months
  Cognitive function will be assessed using the Montreal Cognitive Assessment. The assessment produces a score out of 30. Lower scores indicate increasingly impaired cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Vesna Sossi, Principal Investigator — University of British Columbia
Locations (1):
- Pacific Parkinson's Research Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No